CLINICAL TRIAL: NCT00982839
Title: Rectal Sensory Training - A Randomized Controlled Study of Two Techniques
Brief Title: Rectal Sensory Training - A Study of Two Techniques
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DK057100-08 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Rectal Hyposensitivity; Constipation
MeSH Terms: conditions — Constipation | interventions — Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Syringe Conditioning (Active Comparator): A syringe will be used to inflate the balloon at the end of the probe which is inside of the rectum.
  Interventions: Procedure: Syringe Conditioning
- Barostat Conditioning (Experimental): A barostat machine will be used to inflate the balloon at the end of the probe which is inside of the rectum.
  Interventions: Procedure: Barostat Conditioning

INTERVENTIONS:
Procedure: Syringe Conditioning — A syringe will be used to inflate the balloon at the end of the probe which is inside of the rectum.
  Other Names: Syringe
  Arms: Syringe Conditioning
Procedure: Barostat Conditioning — A barostat machine will be used to inflate the balloon at the end of the probe which is inside of the rectum.
  Other Names: Barostat
  Arms: Barostat Conditioning

SUMMARY:
At least 60% of patients with constipation and dyssynergic defecation (anismus) and between 30-50% of patients with fecal incontinence exhibit impaired rectal sensation. The problem may be improved by biofeedback therapy. Traditionally, biofeedback therapy was performed by using a syringe-assisted technique. Although some respond to this method, many, particularly those with severe rectal hyposensitivity have proved to be refractory. Also, repeated inflation and deflation of a large volume of air, using a hand-held syringe is cumbersome and time consuming. Recently, in pilot observations, the investigators have seen that a barostat-assisted technique of biofeedback therapy was simpler and easier to perform and could possibly be more effective. The investigators' aims are:

1. To perform a randomized controlled study that compares the syringe-assisted sensory conditioning (biofeedback therapy) technique with the barostat assisted sensory conditioning for improving the rectal sensation in patients with rectal hyposensitivity and bowel dysfunction.
2. To investigate the impact of sensory conditioning on psychosocial issues and quality of life.
3. To compare the cost-effectiveness of each therapeutic modality The specific hypotheses that will be tested are;

When compared to those who receive syringe-assisted training, patients receiving barostat training will demonstrate:

1. Lower sensory thresholds for rectal perception (first sensation, desire to defecate and urgency)
2. Greater satisfaction with bowel function (VAS Score), stool frequency,consistency & straining.
3. Better learning ability and greater ease of administering this training.

ELIGIBILITY:
Inclusion Criteria:

* Patients categorized as having dyssynergic defecation or slow transit constipation or normal transit constipation will be eligible.
* All patients must demonstrate rectal hyposensitivity during a manometry with values that are outside 2 S.D. of normal range and demonstrate any two of the following: a) Threshold for 1st sensation > 40 cc. b) Threshold for desire to defecate > 130 cc. c) Threshold for urgency to defecate >180 cc.

Exclusion Criteria:

* Patients taking drugs that are constipating, (e.g.; calcium channel antagonists will either be excluded or drug discontinued).
* Patients with co-morbid illnesses; severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy.
* Neurologic diseases e.g.; head injury, epilepsy, multiple sclerosis, strokes, spinal cord injuries.
* Impaired cognizance (mini mental score of < 15) and/or legally blind.
* Pregnant or likely to conceive during the course of the study. Women with potential for pregnancy must be willing to use contraceptive measures during the study. Urinary pregnancy tests will be performed on such women prior to any radiologic procedures.
* Hirschsprung's disease.
* Alternating constipation and diarrhea (22).
* Ulcerative/Crohns colitis.
* Previous pelvic surgery, rectocele/bladder repair, radical hysterectomy, anal surgery.
* Rectal prolapse or anal fissure. 11) Patients with severe rectal hyposensitivity, first sensation or desire to defecate > 320 cc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2004-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rectal Sensory Thresholds | Trial entry and at the end of 3 months

SECONDARY OUTCOMES:
Satisfaction with bowel function based on Visual Analog Scale (VAS) | Trial Entry and at the end of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, Md, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States